CLINICAL TRIAL: NCT06404723
Title: The Predictive and Prognostic Values of the Fibrinogen to Albumin Ratio and C-reactive Protien to Albumin Ratio in Systemic Lupus Erythematosus Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Manar Gamal Mohamed, Specialist of Physical Medicine, Rheumatology and Rehabilitation at Medical Admintsration at Sohag University, Sohag University
Other Study IDs: soh-Med-24-02-07MD
Record Dates: First submitted 2024-05-05; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, whole blood, plasma, urine sample
  1. Complete blood picture (CBC).
  2. Erythrocyte sedimentation rate (ESR).
  3. C-reactive protein (CRP)
  4. Liver function tests (LFT).
  5. Renal investigations:
     1. Kidney functions
     2. Urine analysis
     3. 24 hours protein in urine and/or A/C ratio or p/c ratio.
     4. eGFR
     5. Renal biopsy.
  6. ANA by IF.
  4. Specific tests:
  1. Fibrinogen to Albumin ratio (FAR).
  2. C-Reactive protein to Albumin Ratio (CAR).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Control Group: : this group contains 50 healthy individual
  Interventions: Diagnostic Test: Fibrinogen to albumin Ratio and C-reactive to Albumin Ratio
- Lupus Simplex (mild to moderate disease) activity Group: this group contains 50 patients with a systemic lupus erythematosus disease activity index 2000 (SLEDAI-2K) score less than 15.
  Interventions: Diagnostic Test: Fibrinogen to albumin Ratio and C-reactive to Albumin Ratio
- Severe disease activity Group: this group contains 50 patients with a systemic lupus erythematosus disease activity index 2000 (SLEDAI-2K) score ≥ 15.
  Interventions: Diagnostic Test: Fibrinogen to albumin Ratio and C-reactive to Albumin Ratio

INTERVENTIONS:
Diagnostic Test: Fibrinogen to albumin Ratio and C-reactive to Albumin Ratio — to detect their relation to disease activity to use as predective and prognostic tools

SUMMARY:
The aim of the study was to study the predictive value of FAR and CAR in order to provide a new predictive biomarkers for the disease activity and prognosis.

DETAILED DESCRIPTION:
A total of 150 participants were included in a Case-Control study:

1. Healthy control group: this group contains 50 healthy individual.
2. Lupus simplex (mild and moderate disease activity) group: this group contains 50 patients with a systemic lupus erythematosus disease activity index 2000 (SLEDAI-2K) score less than 15.
3. Severe disease activity group: this group contains 50 patients with a systemic lupus erythematosus disease activity index 2000 (SLEDAI-2K) score ≥ 15.

Setting:

This study will be conducted to All patients will enter to The Rheumatology Department, Sohag University Hospital for one year.

Inclusion criteria:

Patients diagnosed as SLE according to SLICC 2012 or ACE/EULAR 2017 classification criteria with

1. ≥18 years of age.
2. Complete clinical and laboratory investigations.
3. No concomitant infection, systemic or other autoimmune diseases.

Exclusion criteria:

Patients were excluded from the study if they had any of the following:

1. <18 years of age,
2. Incomplete clinical data and laboratory indicators.
3. End-stage kidney disease (defned as requiring dialysis, kidney transplantation, or estimated glomerular fltration rate (eGFR)<15 mL/min/1.73 m2
4. Patients with:

   1. Acute infectious diseases, HIV infection carriers,
   2. Concomitant systemic diseases such as chronic obstructive lung disease, coronary artery disease, cancer, thyroid function disorder, hematological disorders, acute or chronic liver and renal diseases.
   3. Patients with had other autoimmune diseases, such as rheumatoid arthritis, systemic sclerosis, or primary Sjogren's syndrome.

Methods:

All patients will be subjected to the following:

1. Thorough medical history from the patients
2. Full clinical examination including:

   1. General examination and vital signs.
   2. Complete rheumatological examination.
   3. Systemic lupus erythematosus disease activity index 2000 (SLEDAI-2K) score.
3. Laboratory examinations include:

1. Complete blood picture (CBC). 2. Erythrocyte sedimentation rate (ESR). 3. C-reactive protein (CRP) 4. Liver function tests (LFT). 5. Renal investigations:

1. Kidney functions
2. Urine analysis
3. 24 hours protein in urine and/or A/C ratio or p/c ratio.
4. eGFR
5. Renal biopsy. 6. ANA by IF. 4. Specific tests: a. Fibrinogen to Albumin ratio (FAR). b. C-Reactive protein to Albumin Ratio (CAR).

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed as SLE according to SLICC 2012 or ACE/EULAR 2017 classification criteria with

1. ≥18 years of age.
2. Complete clinical and laboratory investigations.
3. No concomitant infection, systemic or other autoimmune diseases.

Exclusion Criteria:

Patients were excluded from the study if they had any of the following:

1. <18 years of age,
2. Incomplete clinical data and laboratory indicators.
3. End-stage kidney disease (defned as requiring dialysis, kidney transplantation, or estimated glomerular fltration rate (eGFR)<15 mL/min/1.73 m2
4. Patients with:

   1. Acute infectious diseases, HIV infection carriers,
   2. Concomitant systemic diseases such as chronic obstructive lung disease, coronary artery disease, cancer, thyroid function disorder, hematological disorders, acute or chronic liver and renal diseases.
   3. Patients with had other autoimmune diseases, such as rheumatoid arthritis, systemic sclerosis, or primary Sjogren's syndrome.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A total of 150 participants were included in a Case-Control study:
  1. Healthy control group: this group contains 50 healthy individual.
  2. Lupus simplex (mild and moderate disease activity) group: this group contains 50 patients with a systemic lupus erythematosus disease activity index 2000 (SLEDAI-2K) score less than 15.
  3. Severe disease activity group: this group contains 50 patients with a systemic lupus erythematosus disease activity index 2000 (SLEDAI-2K) score ≥ 15.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Fibrinogen/Albumin ratio, C-reactive protein /Albumin ratio | 1-6-2024 to 1-6-2025
  detect if the results approve their use as a predictive and prognostic tools for SLE

IPD SHARING:
Plan to Share IPD: Undecided